CLINICAL TRIAL: NCT07059390
Title: Changi General Hospital Complementary Health Therapy
Brief Title: Concurrent Trials on Nature-Based Therapy for Inpatients in Dementia and Rehabilitation Medicine Wards
Acronym: TGIF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2025-032
Record Dates: First submitted 2025-06-26; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Acquired Brain Injury Including Stroke
Keywords: Dementia; Stroke; Traumatic Brain Injury; Delirium; Nature-Based Therapy
MeSH Terms: conditions — Dementia; Stroke; Brain Injuries, Traumatic; Delirium

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dementia Patients - Intervention (Experimental): Patients with dementia who undergo Nature Immersion Therapy
  Interventions: Behavioral: Nature Immersion Therapy
- Dementia Patients - Control (No Intervention): Patients with dementia who do not undergo Nature Immersion Therapy
- Rehabilitation Patients - Intervention (Experimental): Rehabilitation patients who undergo Nature Immersion Therapy
  Interventions: Behavioral: Nature Immersion Therapy
- Rehabilitation Patients - Control (No Intervention): Rehabilitation patients who do not undergo Nature Immersion Therapy

INTERVENTIONS:
Behavioral: Nature Immersion Therapy — During the length of inpatient stay at Changi General Hospital (CGH), which ranges from 5 to 10 days, the patients and caregivers will be enrolled for a set of 3 nature-based sessions. Each session will be conducted in groups of 4 to 6 patients incorporating a relational multi-sensory experience as well as mind-body connectedness while spending time in nature. Each of the 3 sessions will be 45 minutes each. The nature-based therapy/green social prescription plan will be conducted in groups guided by a trained CGH staff (Allied Health Professionals/Nurse). This Green social prescribing plan (Playbook) will be integrated into inpatient's care plan. Caregivers of the enrolled patients will also be part of the therapy group following the necessary consent.
  Arms: Dementia Patients - Intervention; Rehabilitation Patients - Intervention

SUMMARY:
Nature-based Therapy, such as forest bathing and horticultural therapy, has been shown to have physical, psychological and emotional health benefits. We posit that personalised and guided Nature-based Therapy, which leverages the benefits of therapeutic gardens in an urban hospital setting, improves the overall wellbeing of elderly inpatients with dementia (aged >65 years old) and their caregivers, as well as patients undergoing inpatient rehabilitation. To determine the effectiveness of Nature-based Therapy for these two inpatient populations, we designed a pilot study, TGIF, to be conducted at the dementia and rehabilitation medicine wards at Changi General Hospital in Singapore.

DETAILED DESCRIPTION:
TGIF consists of two concurrent trials targeting two patient populations: elderly inpatients with dementia admitted to the dementia ward, and inpatients undergoing inpatient rehabilitation at the rehabilitation wards in a tertiary teaching hospital in Singapore. At the dementia wards, we aim to determine if Nature-based Therapy improved the neuropsychiatric symptoms such as agitation, restlessness and aggression among elderly inpatients living with cognitive impairment, defined as either delirium or dementia or both. Concurrent with the improved neuropsychiatric symptoms, the study team will also study the improved quality of life among the family, caregivers and hence reduced caregiver burden. At the rehabilitation medicine wards, we aim to determine if Nature-based Therapy improves mood, physical function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients with dementia:

1. Age 65-100 years old
2. Have a diagnosis of delirium/ dementia or both.
3. Have diagnosis of dementia with and without behavioural symptoms of dementia (BPSD)
4. Ability to communicate with the Nature-based Therapist (in languages such as English, Mandarin Chinese, Chinese dialects or Malay)
5. Manageable behavioural symptoms and able to focus attention for minimum of 30 minutes

Rehabilitation Medicine patients:

1. Age 21-100 years old
2. Acquired brain injury with residual impairments, which can be either in the i) motor, and/or ii) cognitive domains, and/or iii) suspected or diagnosed mood disorders (including adjustment disorder, depression and anxiety disorders) -patients would then be stratified according to the category(s) of impairments both for consideration of interventions and for outcome measures/analysis
3. Additional Physical/Cognitive Criteria required will depend on range of specific therapeutic activities that could be prescribed/administered (eg.at least 1 upper limb with Manual Muscle Testing (MMT) of at least 3/5, with ability for active grasp/release, ability to sustain attention for the duration of the session, cognitive Functional Independence Measure (FIM) score of at least 25 points etc)

Exclusion Criteria:

1. In isolation due to contact, droplet or airborne precautions
2. Unable to provide consent and lack of surrogate decision maker to provide consent
3. Poorly managed psychiatric or behaviour symptoms with threats to others surrounding them.
4. Age < 21 years
5. Patients who are haemodynamically unstable.
6. Patients on strict bed rest

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Pittsburg Agitation Scale | Baseline and at the end of intervention, an average 7 days
  The Pittsburgh Agitation Scale (PAS) is a quick, observational tool used to assess the severity of agitation in dementia patients, focusing on four behavioral dimensions: aberrant vocalizations, motor agitation, aggressiveness, and resistance to care
DASS-21 | Baseline and at the end of intervention, an average of 7 days
  The DASS-21 (Depression, Anxiety, and Stress Scale - 21 Items) is a self-report questionnaire designed to measure the severity of symptoms related to depression, anxiety, and stress in adults. It consists of 21 questions, with seven questions for each of the three scales: depression, anxiety, and stress.

SECONDARY OUTCOMES:
EQ-5D-5L | Baseline and at the end of intervention, an average of 7 days
  The EQ-5D-5L is a generic, self-completed questionnaire that assesses health-related quality of life (HRQoL) across five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with five levels of severity for each dimension, and includes a visual analogue scale (EQ VAS).
Zarit Burden Interview | Baseline and at the end of intervention, an average of 7 days
  The Zarit Burden Interview (ZBI) is a widely used tool to assess the level of caregiver burden experienced by individuals who care for people with chronic illnesses. It is a self-report questionnaire that evaluates the physical, emotional, and social impact of caregiving on the caregiver's well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Si Ching Lim, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The dataset is restricted due to ethical limitations.

REFERENCES:
- [Background] Hansen MM, Jones R, Tocchini K. Shinrin-Yoku (Forest Bathing) and Nature Therapy: A State-of-the-Art Review. Int J Environ Res Public Health. 2017 Jul 28;14(8):851. doi: 10.3390/ijerph14080851. PMID 28788101
- [Background] Vibholm AP, Christensen JR, Pallesen H. Nature-based rehabilitation for adults with acquired brain injury: a scoping review. Int J Environ Health Res. 2020 Dec;30(6):661-676. doi: 10.1080/09603123.2019.1620183. Epub 2019 May 27. PMID 31131619
- [Background] Ng KST, Sia A, Ng MKW, Tan CTY, Chan HY, Tan CH, Rawtaer I, Feng L, Mahendran R, Larbi A, Kua EH, Ho RCM. Effects of Horticultural Therapy on Asian Older Adults: A Randomized Controlled Trial. Int J Environ Res Public Health. 2018 Aug 9;15(8):1705. doi: 10.3390/ijerph15081705. PMID 30096932
- [Background] Howarth M, Brettle A, Hardman M, Maden M. What is the evidence for the impact of gardens and gardening on health and well-being: a scoping review and evidence-based logic model to guide healthcare strategy decision making on the use of gardening approaches as a social prescription. BMJ Open. 2020 Jul 19;10(7):e036923. doi: 10.1136/bmjopen-2020-036923. PMID 32690529
- [Background] Antonelli M, Barbieri G, Donelli D. Effects of forest bathing (shinrin-yoku) on levels of cortisol as a stress biomarker: a systematic review and meta-analysis. Int J Biometeorol. 2019 Aug;63(8):1117-1134. doi: 10.1007/s00484-019-01717-x. Epub 2019 Apr 18. PMID 31001682
- [Background] Li Q. Effect of forest bathing trips on human immune function. Environ Health Prev Med. 2010 Jan;15(1):9-17. doi: 10.1007/s12199-008-0068-3. PMID 19568839
- [Background] Siah CJR, Goh YS, Lee J, Poon SN, Ow Yong JQY, Tam WW. The effects of forest bathing on psychological well-being: A systematic review and meta-analysis. Int J Ment Health Nurs. 2023 Aug;32(4):1038-1054. doi: 10.1111/inm.13131. Epub 2023 Mar 2. PMID 36864583
- [Background] Kavanaugh J, Hardison ME, Rogers HH, White C, Gross J. Assessing the Impact of a Shinrin-Yoku (Forest Bathing) Intervention on Physician/Healthcare Professional Burnout: A Randomized, Controlled Trial. Int J Environ Res Public Health. 2022 Nov 4;19(21):14505. doi: 10.3390/ijerph192114505. PMID 36361384